CLINICAL TRIAL: NCT03081481
Title: Multi-Centre, Ph IIb Study, Evaluating Safety & Efficacy of Targeted Intraprostatic Admin of PRX302 to Treat Men With Histologically Proven, Clinically Significant, Localised Prostate Cancer Associated With MRI Lesion
Brief Title: Intraprostatic PRX302 Injection to Treat Localised Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sophiris Bio Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRX302-2-08
Record Dates: First submitted 2017-03-07; First posted 2017-03-16 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer
Keywords: Intraprostatic; MRI lesion; Prostate biopsies
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PRX302

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRX302 (Experimental): intraprostatic administration
  Interventions: Drug: PRX302

INTERVENTIONS:
Drug: PRX302 — Single prostate cancer lesion injected with PRX302
  Other Names: Topsalysin

SUMMARY:
The purpose of this study is to determine a safe, effective, and tolerable dose of PRX302 for the treatment of low to intermediate risk prostate cancer.

DETAILED DESCRIPTION:
A multi-centre, open label, phase IIb study, evaluating the safety, tolerability and efficacy of a targeted intraprostatic focal administration in development. The study will treat approximately 40 men who meet the eligibility criteria, and give written consent. Safety and tolerability will be assessed post-treatment over 26 weeks. Efficacy will be assessed by biopsy and imaging (mpMRI) at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy ≥ 10 years.
* Serum prostate-specific antigen (PSA) ≤ 15ng/mL.
* A histologically proven, clinically significant lesion visible on mpMRI (magnetic resonance imaging) that is accessible to PRX302 transperineal injection.
* Radiological stage T1-T2 N0 Mx/M0 disease.
* Targeted prostate biopsy within 6 months prior to dosing, with a clinically significant lesion correlating with an mpMRI visible lesion.

Exclusion Criteria:

* Previous radiation therapy to the pelvis.
* Androgen suppression or anti-androgen therapy within the 12 months prior to dosing, for prostate cancer.
* Use of 5-alpha reductase inhibitor within the 3 months prior to dosing.
* Evidence of metastatic disease or nodal disease outside the prostate on bone scan or cross-sectional imaging.
* Inability to tolerate transrectal ultrasound (TRUS).
* Known allergy to latex or gadolinium (Gd).
* Prior rectal surgery preventing insertion of the TRUS probe.
* Any previous ablative procedures performed on the prostate, e.g., electroporation, radiofrequency ablation, high-intensity focused ultrasound (HIFU), cryosurgery, photochemical, thermal or microwave therapy to treat cancer of the prostate.
* Unable to have pelvic MRI scanning (severe claustrophobia, permanent cardiac pacemaker, metallic implant, etc., likely to contribute significant artifact to images).

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 26 weeks post administration
  Treatment-emergent adverse events (TEAEs), including both serious and non-serious AEs, and assessments of severity and relatedness to both the study drug agent (PRX302) and the rest of the injection procedure

SECONDARY OUTCOMES:
Proportion of patients with an absence of clinically significant prostate cancer in the targeted area at 24 weeks post-administration of PRX302, as determined by a transperineal targeted biopsy [Efficacy] | 24 weeks post administration
  Clinically significant disease is defined as Gleason 7, or in the presence of Gleason 3+3 a maximum cancer core length > 6 mm

CONTACTS AND LOCATIONS:
Overall Officials: Hashim U Ahmed, MD, Principal Investigator — Imperial College London
Locations (8):
- United States (4):
  - Vantage Health, Ocala, Florida
  - Chesapeake Urology Associates, Baltimore, Maryland
  - New York Urology Associates, New York, New York
  - Baylor Scott & White Memorial Hospital and Clinic, Temple, Texas
- United Kingdom (4):
  - Princess Alexandra Hospital, Harlow
  - Imperial College, London
  - University College Hospital (UCLH), London
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No